CLINICAL TRIAL: NCT06714279
Title: Laparoscopic-Assisted Transversus Abdominus Plane Block Versus Intraperitoneal Irrigation of Local Anesthetic for Patients Undergoing Laparoscopic Cholecystectomy - A Prospective, Randomised Clinical Trial
Brief Title: Laparoscopic-Assisted Transversus Abdominus Plane Block Versus Intraperitoneal Irrigation of Local Anesthetic for Patients Undergoing Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Matthew Davey, Specialist Registrar in General Surgery, Royal College of Surgeons, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24.71
Record Dates: First submitted 2024-11-23; First posted 2024-12-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Cholecystectomy; TAP Block; Local Anesthetic
Keywords: Laparoscopic cholecystectomy; TAP block; Transversus abdominus plane block; Local anesthetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group - Tap Block (Other): Study Group: Study group: Laparoscopic Transversus Abdominis Plane in four points: above the umbilicus on the left side; dose calculation 2.5mg per body weight.
  After the cholecystectomy is done and just before withdrawing port and deflating the abdomen, the operating surgeon will advance a needle into the abdominal wall to the level of the preperitoneal space. Once the needle tip is seen, it is withdrawn slowly and gently about 0.5cm above/superficial to the transversus abdominis (TA) muscle. The surgeon then infiltrates the local anaesthetic into the plane, and the right plane is confirmed by visualising a uniform protrusion downwards of the TA muscle fibres (Doyle's bulge). Seeing a preperitoneal or muscle blister laparoscopically indicates that the infiltration is deeper to this plane, and the needle should be withdrawn more superficially.
  Interventions: Drug: Tap Block - Bupivacaine
- Control Group - Intraperitoneal Local Anesthetic onto Liver (Placebo Comparator): Administration of local anesthetic to the liver using, dose calculation 2.5mg per body weight.
  Interventions: Drug: Intraperitoneal infiltration to liver

INTERVENTIONS:
Drug: Tap Block - Bupivacaine — The medicinal product for both groups is the same - Bupivacaine. The mode of administration is what this study is reviewing: Control group (Intraperitoneal infiltration to liver) and Study Group - Laparoscopic Transversus Abdominis Plane Block (LTap Block)
  Arms: Study Group - Tap Block
Drug: Intraperitoneal infiltration to liver — The medicinal product for both groups is the same - Bupivacaine. The mode of administration is what this study is reviewing: Control group (Intraperitoneal infiltration to liver) and Study Group - Laparoscopic Transversus Abdominis Plane Block (LTap Block)
  Arms: Control Group - Intraperitoneal Local Anesthetic onto Liver

SUMMARY:
This study is being performed to investigate whether the administration of local anaesthetic into the muscles in the abdomen or onto squirting the local anaesthetic onto the liver following keyhole gallbladder surgery is more beneficial in reducing pain post-operatively.

Keyhole gallbladder surgery is typically performed under general anaesthesia (or while the patient is 'fully asleep'), however doctors use other pain relief types to reduce pain after the operation. One of these options is local anaesthetic, which involves the injection of an medication into or onto the part of the body which has been operated on. The reason for doing this is to reduce the pain felt by the patient in the part if the body where the operation occurred. The best way of using these medications remain unclear.

The local anaesthetic being used in the study is fully approved for use in Ireland and the drug itself is not being tested. In other words, the drug is not an experimental drug. Local anaesthetic drugs are given in different ways in patients who have just had the keyhole surgery on their gall bladder (this is the surgery that you are about to have).

Therefore, the aim of this study is to compare two ways of giving patients these local anaesthetic medications following key-hole gallbladder surgery. These include (1) injecting the medication into the skin at the surgical wounds and squirting it onto the liver (where the gallbladder has been removed from), or (2) injecting the medication into the skin at the surgical wounds and into the muscles in the abdomen (known formally as a transversus abdominus plane block).

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy remains the cornerstone in treating benign diseases of the gallbladder and biliary tree, with approximately 5,000 of these procedures being performed annually in the Republic of Ireland. While significant complications, including bile leak, common bile duct injury (CBDI), and converting to an open incision, are typically discussed in detail when counselling patients in the preoperative setting, post-operative pain in the first 24-hours after surgery remains the main barrier of early discharge following the procedure. To counteract this issue, multimodal analgesic strategies have practically been adopted to minimise post-operative pain following laparoscopic cholecystectomy, as outlined by the Procedure Specific Post-Operative Pain Management (PROSPECT) in their review and recommendations. More specifically, the PROSPECT guidelines provide GRADE A recommendations in support of both standard paracetamol and non-steroidal anti-inflammatory (or cyclooxygenase-2 specific inhibitors), combined with surgical site local anaesthetic infiltration in patients in the peri-operative setting 'as the first line for routine use'.

Despite these recommendations, there remains ambiguity in the surgical literature surrounding to the optimal strategy for the infiltration of local anaesthetic; previous data has coherently demonstrated the superiority of surgical site wound infiltration, intraperitoneal infiltration and intra-abdominal wall blocks with local anaesthetic agents in reducing post-operative pain relative to placebo. In particular, data from a previous randomised clinical trial (RCT) has indicated that infiltrating the gallbladder fossa with local anaesthetic is more effective in reducing post-operative pain than local wound infiltration, however these results were subsequently refuted in a sequential RCT, leaving ambiguity as to the effect of this technique in reducing post-operative pain. Furthermore, recent RCTs have demonstrated that infiltration of local anaesthetic into either transversus abdominus plane (TAP) or the rectus sheath intraoperatively reduced post-operative pain compared to infiltration into the wound alone, directly reducing the post-operative morphine requirement. While ultrasound-guided transversus abdominus plane (US-TAP) are now commonly utilised in the perioperative setting following laparoscopic cholecystectomy, the suitability of a laparoscopic-guided approach (L-TAP) has been less well established within the surgical literature.

Given the contrasting results of these previous studies, there remains no consensus as to the validity of using L-TAP or intraperitoneal infiltration of local anaesthetic to the liver bed as contemporary modes of delivering local anaesthetic following laparoscopic cholecystectomy. Accordingly, the aim of this study was to perform a prospective, randomised study evaluating the benefit of L-TAP or intraperitoneal infiltration in patients indicated to undergo laparoscopic cholecystectomy. This study is a parallel two-arm study which will evaluate outcomes following local anesthetic infiltration (1) directly into the laparoscopic port sites combined with intraperitoneal infiltration, and (2) directly into the laparoscopic port sites combined with laparoscopic infiltration via TAP block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older will be considered for recruitment into this study if they are indicated to undergo elective laparoscopic cholecystectomy

Exclusion Criteria:

* Patients failing to meet the above inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Post operative pain measured via Visual Anaolgue Scores | 1-hour, 3-hours, 6-hours, 12-hours and 24-hours
  The primary objective for the study is to quantify and analyse differences in the post-operative resting and shoulder tip pain as measured using VAS at 1-hour, 3-hours, 6-hours, 12-hours and 24-hours following laparoscopic cholecystectomy. Thereafter, the further opioid analgesic requirements for each patient will be recorded for the duration of their inpatient stay and also the total sum of opioids prescribed for these patients on discharge (measured using morphine equivalents).

CONTACTS AND LOCATIONS:
Overall Officials: Arnold DK Hill, MB MCh FRCS, Principal Investigator — RCSI
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided